CLINICAL TRIAL: NCT00329550
Title: A 26-week, Multi-center, Open-label Study to Investigate the Efficacy and Safety of CDP870 in Active Crohn's Disease Patients, Who Showed Clinical Efficacy in a Remission Induction Study (Study C87037 [NCT00291668]), at Week 26 After Subcutaneous Administration of CDP870 400 mg From Week 8 Until Week 24 at 4-week Intervals
Brief Title: Maintenance Study of Certolizumab Pegol (CZP) in Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87047; 2014-004354-34 (EudraCT Number)
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2009-11-10 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-02

CONDITIONS: Crohn's Disease
Keywords: Certolizumab pegol; Cimzia; CZP
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CZP 400 mg / Placebo (Experimental): Certolizumab pegol (CZP) 400 mg in this extension study / Placebo in double-blind main study (NCT00291668)
  Interventions: Biological: Certolizumab pegol (CZP)
- CZP 400 mg / CZP 200 mg (Experimental): Certolizumab pegol (CZP) 400 mg in this extension study / Certolizumab pegol (CZP) 200 mg in double-blind main study (NCT00291668)
  Interventions: Biological: Certolizumab pegol (CZP)
- CZP 400 mg / CZP 400 mg (Experimental): Certolizumab pegol (CZP) 400 mg in this extension study / Certolizumab pegol (CZP) 400 mg in double-blind main study (NCT00291668)
  Interventions: Biological: Certolizumab pegol (CZP)

INTERVENTIONS:
Biological: Certolizumab pegol (CZP) — Certolizumab pegol (CZP) 400 mg administered subcutaneously in a liquid formulation at Weeks 8, 12, 16, 20 and 24 relative to the start of the 6-week double-blind main study C87037 (NCT00291668) where subjects received Placebo at Weeks 0, 2 and 4.
  Other Names: CDP870; Cimzia; CZP
  Arms: CZP 400 mg / Placebo
Biological: Certolizumab pegol (CZP) — Certolizumab pegol (CZP) 400 mg administered subcutaneously in a liquid formulation at Weeks 8, 12, 16, 20 and 24 relative to the start of the 6-week double-blind main study C87037 (NCT00291668) where subjects received certolizumab pegol (CZP) 200 mg at Weeks 0, 2 and 4.
  Other Names: CDP870; Cimzia; CZP
  Arms: CZP 400 mg / CZP 200 mg
Biological: Certolizumab pegol (CZP) — Certolizumab pegol (CZP) 400 mg administered subcutaneously in a liquid formulation at Weeks 8, 12, 16, 20 and 24 relative to the start of the 6-week double-blind main study C87037 (NCT00291668) where subjects received certolizumab pegol 400 mg at Weeks 0, 2 and 4.
  Other Names: CDP870; Cimzia; CZP
  Arms: CZP 400 mg / CZP 400 mg

SUMMARY:
This is a multi-centre, open-label extension study in subjects who showed clinical response to induction therapy in the treatment of subjects with active Crohn's disease in the double-blind main study C87037 (NCT00291668).

DETAILED DESCRIPTION:
In the double-blind main study subjects were dosed at Weeks 0, 2 and 4, with the primary outcome, clinical response, being assessed at Week 6. Subjects who showed clinical response at Week 6 were eligible to enter this open-label extension study. The first visit in this extension study was 2 weeks after Week 6, i.e., Week 8. Subjects in this extension study were dosed at Weeks 8, 12, 16, 20 and 24, with the primary outcome, clinical response, being assessed at Week 26. All week numbers quoted are relative to the start of the double-blind main study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in main double-blind induction study C87037 (NCT00291668) and showed clinical efficacy

Exclusion Criteria:

* Subjects who experienced aggravation of Crohn's disease during main double-blind induction study C87037 (NCT00291668) and required treatment change

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Principal Investigator — +1 877 822 9493 (UCB)
Locations (23):
- Japan (23):
  - Aichi-Gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Toyohashi, Aichi-ken
  - Kashiwa, Chiba
  - Sakura, Chiba
  - Chikusino, Fukuoka
  - Fukuoka, Fukuoka
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Kagoshima, Kagoshima-ken
  - Yokohama, Kanagawa
  - Miyazaki-Gun, Miyazaki
  - Nagasaki, Nagasaki
  - Niigata, Niigata
  - Kurashiki, Okayama-ken
  - Tyuto-gun, Okinawa
  - Osaka, Osaka
  - Suita, Osaka
  - Ōtsu, Shiga
  - Shinjyuku/Tokyo, Tokyo
  - Shinjyuku, Tokyo

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment into this extension study was between March 2006 and April 2008. Of the 26 hospitals and medical centers throughout Japan in the main study, 16 sites went on to enter subjects in this extension study.
Pre-assignment Details: To enter this single-group extension study, C87047 (NCT00329550), subjects had to have responded at Week 6 of the double-blind main study, C87037 (NCT00291668). Recruitment details are provided for the 40 subjects who entered this extension study by the three possible treatment sequences received across both studies.
Groups:
- CZP 400 mg / Placebo: Certolizumab pegol (CZP) 400 mg (5 doses 4-weekly) in this extension study / Placebo (3 doses 2-weekly) in the 6-week double-blind main study (NCT00291668)
- CZP 400 mg / CZP 200 mg: Certolizumab pegol (CZP) 400 mg (5 doses 4-weekly) in this extension study / Certolizumab pegol (CZP) 200 mg (3 doses 2-weekly) in the 6-week double-blind main study (NCT00291668)
- CZP 400 mg / CZP 400 mg: Certolizumab pegol (CZP) 400 mg (5 doses 4-weekly) in this extension study / Certolizumab pegol (CZP) 400 mg (3 doses 2-weekly) in the 6-week double-blind main study (NCT00291668)
Period: Overall Study
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Started | 9 | 15 | 16 (1 subject in Safety Set is not in Full Analysis Set due to Good Clinical Practice non-compliance.)
Completed | 5 | 11 | 12
Not Completed | 4 | 4 | 4
Not completed — Adverse Event | 3 | 4 | 2
Not completed — Withdrawal of Consent | 1 | 0 | 1
Not completed — Due to Relocation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg | Total
Number analyzed (Participants) | 9 | 15 | 16 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 2 | 6.0
  Between 18 and 65 years | 8 | 12 | 14 | 34.0
  >=65 years | 0 | 0 | 0 | 0.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (10.4) | 29.3 (9.1) | 33.3 (10.0) | 31.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 9.0
  Male | 7 | 12 | 12 | 31.0
Region of Enrollment [Number; unit: participants]
  Japan | 9 | 15 | 16 | 40.0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 26
Description: CDAI responders are subjects achieving either clinical response (a reduction in CDAI score of ≥100 points from Week 0), or remission (CDAI ≤150). CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: Week 0 and Week 26 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 26' is 18 weeks after the first visit in this extension study.
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). All 39 subjects in the Full Analysis Set (FAS) were included in this summary. If a subject withdrew or received rescue therapy, they were counted as a non-responder in that study from that time-point onwards.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 44.4 | 73.3 | 60.0
  Percentage of CDAI non-responders | 55.6 | 26.7 | 40.0

2. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 8
Description: CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 0 and Week 8 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 8' is the first visit in this extension study.
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). Subjects in the Full Analysis Set (FAS) with data at both time-points are included. Data collected after receipt of rescue therapy have been set to missing in that study. [Week 8 is the start of Study C87047].
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
score on a scale | -126.7 (100.9) | -124.9 (76.7) | -141.8 (62.4)

3. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 12
Description: as for outcome 2
Time Frame: Week 0 and Week 12 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 12' is 4 weeks after the first visit in this extension study.
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). Subjects in the Full Analysis Set (FAS) with data at both time-points are included. Data collected after receipt of rescue therapy in a study have been set to missing in that study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
score on a scale | -152.6 (96.8) | -145.4 (80.5) | -152.8 (54.7)

4. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 16
Description: as for outcome 2
Time Frame: Week 0 and Week 16 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 16' is 8 weeks after the first visit in this extension study.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
score on a scale | -162.8 (98.9) | -142.2 (84.3) | -143.3 (69.6)

5. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 20
Description: as for outcome 2
Time Frame: Week 0 and Week 20 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 20' is 12 weeks after the first visit in this extension study.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
score on a scale | -147.0 (38.8) | -149.4 (85.6) | -130.7 (70.1)

6. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 24
Description: as for outcome 2
Time Frame: Week 0 and Week 24 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 24' is 16 weeks after the first visit in this extension study.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
score on a scale | -158.6 (53.7) | -153.3 (53.7) | -138.9 (80.0)

7. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Week 26
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
score on a scale | -131.1 (32.8) | -173.8 (46.5) | -153.1 (70.8)

8. Secondary Outcome: Change From Week 0 in Crohn's Disease Activity Index (CDAI) Score at Last Visit [Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals]
Description: as for outcome 2
Time Frame: Week 0 and Last Visit (Week 26 relative to the start of the 6-week double-blind main study (NCT00291668) for completers or the Withdrawal Visit for premature withdrawals). 'Week 26' is 18 weeks after the first visit in this extension study.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
score on a scale | -132.7 (62.6) | -143.2 (88.5) | -152.5 (67.9)

9. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 8
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 55.6 | 66.7 | 80.0
  Percentage of CDAI non-responders | 44.4 | 33.3 | 20.0

10. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 12
Description: as for outcome 1
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 77.8 | 73.3 | 86.7
  Percentage of CDAI non-responders | 22.2 | 26.7 | 13.3

11. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 16
Description: as for outcome 1
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 77.8 | 60.0 | 66.7
  Percentage of CDAI non-responders | 22.2 | 40.0 | 33.3

12. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 20
Description: as for outcome 1
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 66.7 | 60.0 | 60.0
  Percentage of CDAI non-responders | 33.3 | 40.0 | 40.0

13. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 24
Description: as for outcome 1
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 44.4 | 60.0 | 53.3
  Percentage of CDAI non-responders | 55.6 | 40.0 | 46.7

14. Secondary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Last Visit [Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals]
Description: as for outcome 1
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of CDAI responders | 44.4 | 73.3 | 60.0
  Percentage of CDAI non-responders | 55.6 | 26.7 | 40.0

15. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 8
Description: The Crohn's Disease Activity Index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A CDAI score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: Week 8 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 8' is the first visit in this extension study.
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). All 39 subjects in the Full Analysis Set (FAS) were included in this summary. If a subject withdrew or received rescue therapy, they were counted as not in remission in that study from that time-point onwards.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 33.3 | 40.0 | 53.3
  Percentage of subjects not in remission | 66.7 | 60.0 | 46.7

16. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 12
Description: as for outcome 15
Time Frame: Week 12 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 12' is 4 weeks after the first visit in this extension study.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 44.4 | 46.7 | 53.3
  Percentage of subjects not in remission | 55.6 | 53.3 | 46.7

17. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 16
Description: as for outcome 15
Time Frame: Week 16 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 16' is 8 weeks after the first visit in this extension study.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 44.4 | 46.7 | 40.0
  Percentage of subjects not in remission | 55.6 | 53.3 | 60.0

18. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 20
Description: as for outcome 15
Time Frame: Week 20 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 20' is 12 weeks after the first visit in this extension study.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 22.2 | 53.3 | 40.0
  Percentage of subjects not in remission | 77.8 | 46.7 | 60.0

19. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 24
Description: as for outcome 15
Time Frame: Week 24 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 24' is 16 weeks after the first visit in this extension study.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 22.2 | 46.7 | 40.0
  Percentage of subjects not in remission | 77.8 | 53.3 | 60.0

20. Secondary Outcome: Percentage of Subjects Achieving Remission at Week 26
Description: as for outcome 15
Time Frame: Week 26 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 26' is 18 weeks after the first visit in this extension study.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 22.2 | 46.7 | 46.7
  Percentage of subjects not in remission | 77.8 | 53.3 | 53.3

21. Secondary Outcome: Percentage of Subjects Achieving Remission at Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals)
Description: as for outcome 15
Time Frame: Last Visit (Week 26 relative to the start of the 6-week double-blind main study (NCT00291668) for completers or the Withdrawal Visit for premature withdrawals). 'Week 26' is 18 weeks after the first visit in this extension study.
Population: as for outcome 15
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of subjects in remission | 22.2 | 46.7 | 46.7
  Percentage of subjects not in remission | 77.8 | 53.3 | 53.3

22. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the earliest of:
  * time to an increase from Week 6 of ≥100 points in Crohn's Disease Activity Index (CDAI) score and CDAI >175 points for at least 2 consecutive visits,
  * time to use of rescue therapy, or,
  * time to subject withdrawal from the study.
Time Frame: Week 6 to Week 26 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 6' is the last visit in the double-blind main study and 'Week 26' is 18 weeks after the first visit in this extension study.
Population: Responders at Week 6 of Study C87037 (NCT00291668) could enter this extension study C87047 (NCT00329550). As so few subjects experienced disease progression in this study it was not possible to calculate the median time to disease progression. Please see post-hoc outcome measure 80 where the number of subjects with disease progression is presented.
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Change From Week 0 to Week 8 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: The IBDQ Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
score on a scale | 33.8 (25.6) | 30.4 (25.8) | 23.7 (20.3)

24. Secondary Outcome: Change From Week 0 to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: as for outcome 23
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
score on a scale | 37.6 (27.0) | 29.9 (28.6) | 25.5 (20.3)

25. Secondary Outcome: Change From Week 0 to Week 16 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: as for outcome 23
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
score on a scale | 31.0 (31.6) | 30.1 (25.4) | 22.6 (22.4)

26. Secondary Outcome: Change From Week 0 to Week 20 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: as for outcome 23
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
score on a scale | 32.2 (20.7) | 31.6 (27.6) | 19.2 (25.9)

27. Secondary Outcome: Change From Week 0 to Week 24 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: as for outcome 23
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
score on a scale | 34.0 (13.4) | 32.7 (24.6) | 23.6 (22.5)

28. Secondary Outcome: Change From Week 0 to Week 26 in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: as for outcome 23
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
score on a scale | 33.4 (17.0) | 38.4 (27.0) | 28.2 (19.5)

29. Secondary Outcome: Change From Week 0 to Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) in Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Global Score is the sum of 32 responses, each ranging from 0 to 7, thus the Global Score ranges from 0 to 224; a higher score indicating a better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
score on a scale | 28.0 (21.5) | 33.3 (27.7) | 26.1 (20.1)

30. Secondary Outcome: Change From Week 0 to Week 8 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: The IBDQ Bowel Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
score on a scale | 10.7 (5.8) | 10.3 (8.6) | 9.5 (10.2)

31. Secondary Outcome: Change From Week 0 to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: as for outcome 30
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
score on a scale | 12.6 (6.9) | 10.2 (10.8) | 9.8 (8.5)

32. Secondary Outcome: Change From Week 0 to Week 16 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: as for outcome 30
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
score on a scale | 9.9 (8.3) | 8.8 (9.6) | 6.7 (7.2)

33. Secondary Outcome: Change From Week 0 to Week 20 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: as for outcome 30
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
score on a scale | 9.5 (8.3) | 11.3 (9.7) | 6.7 (8.8)

34. Secondary Outcome: Change From Week 0 to Week 24 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: as for outcome 30
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
score on a scale | 11.0 (3.0) | 10.4 (8.7) | 8.0 (9.5)

35. Secondary Outcome: Change From Week 0 to Week 26 in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: as for outcome 30
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
score on a scale | 11.6 (4.2) | 12.0 (10.4) | 8.8 (9.9)

36. Secondary Outcome: Change From Week 0 to Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) in Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Bowel Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
score on a scale | 9.6 (5.8) | 10.7 (10.1) | 8.1 (9.8)

37. Secondary Outcome: Change From Week 0 to Week 8 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: The IBDQ Systemic Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
score on a scale | 7.6 (7.0) | 7.1 (5.9) | 5.7 (4.7)

38. Secondary Outcome: Change From Week 0 to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: as for outcome 37
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
score on a scale | 7.4 (7.8) | 7.4 (6.0) | 5.9 (5.4)

39. Secondary Outcome: Change From Week 0 to Week 16 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: as for outcome 37
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
score on a scale | 6.8 (9.1) | 7.9 (5.9) | 5.9 (6.5)

40. Secondary Outcome: Change From Week 0 to Week 20 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: as for outcome 37
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
score on a scale | 7.5 (3.4) | 7.3 (6.6) | 4.9 (6.2)

41. Secondary Outcome: Change From Week 0 to Week 24 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: as for outcome 37
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
score on a scale | 8.2 (3.1) | 7.5 (6.7) | 6.2 (3.5)

42. Secondary Outcome: Change From Week 0 to Week 26 in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: as for outcome 37
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
score on a scale | 6.4 (3.5) | 8.7 (5.6) | 7.2 (3.6)

43. Secondary Outcome: Change From Week 0 to Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) in Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Systemic Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
score on a scale | 5.1 (6.8) | 8.8 (5.1) | 7.2 (3.4)

44. Secondary Outcome: Change From Week 0 to Week 8 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: The IBDQ Emotional Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
score on a scale | 9.4 (7.0) | 7.5 (8.6) | 5.1 (8.7)

45. Secondary Outcome: Change From Week 0 to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: as for outcome 44
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
score on a scale | 10.8 (7.6) | 7.7 (8.2) | 5.4 (9.6)

46. Secondary Outcome: Change From Week 0 to Week 16 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: as for outcome 44
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
score on a scale | 8.0 (8.2) | 7.8 (8.4) | 6.1 (9.6)

47. Secondary Outcome: Change From Week 0 to Week 20 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: as for outcome 44
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
score on a scale | 8.5 (9.4) | 6.8 (9.4) | 4.1 (10.3)

48. Secondary Outcome: Change From Week 0 to Week 24 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: as for outcome 44
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
score on a scale | 8.3 (6.1) | 8.6 (9.1) | 6.2 (10.3)

49. Secondary Outcome: Change From Week 0 to Week 26 in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: as for outcome 44
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
score on a scale | 9.4 (7.2) | 11.3 (11.1) | 6.8 (8.6)

50. Secondary Outcome: Change From Week 0 to Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) in Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Emotional Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
score on a scale | 7.4 (6.8) | 9.0 (11.6) | 5.8 (9.0)

51. Secondary Outcome: Change From Week 0 to Week 8 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: The IBDQ Social Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
score on a scale | 6.1 (7.4) | 5.5 (7.1) | 3.5 (4.0)

52. Secondary Outcome: Change From Week 0 to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: as for outcome 51
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
score on a scale | 6.9 (7.9) | 4.5 (8.9) | 4.5 (4.1)

53. Secondary Outcome: Change From Week 0 to Week 16 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: as for outcome 51
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
score on a scale | 6.4 (7.7) | 5.6 (7.3) | 4.0 (4.2)

54. Secondary Outcome: Change From Week 0 to Week 20 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: as for outcome 51
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
score on a scale | 6.7 (5.8) | 6.1 (7.9) | 3.6 (5.9)

55. Secondary Outcome: Change From Week 0 to Week 24 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: as for outcome 51
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
score on a scale | 6.5 (6.1) | 6.2 (7.8) | 3.3 (4.3)

56. Secondary Outcome: Change From Week 0 to Week 26 in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: as for outcome 51
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
score on a scale | 6.0 (5.8) | 6.4 (7.8) | 5.7 (5.2)

57. Secondary Outcome: Change From Week 0 to Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) in Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) Social Domain Sub-Score is the sum of 8 responses, each ranging from 0 to 7, thus the Sub-Score ranges from 0 to 56; a higher score indicating a better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
score on a scale | 5.9 (6.0) | 4.8 (8.5) | 5.2 (5.2)

58. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 0
Time Frame: Week 0 (relative to the start of the 6-week double-blind main study (NCT00291668)). 'Week 0' is the Baseline visit in the double-blind main study.
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). Subjects in the Full Analysis Set (FAS) with data at this time-point are included. Data collected after receipt of rescue therapy in a study have been set to missing in that study.
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
mg/L | 21.37 [1.0 to 68.0] | 26.31 [11.0 to 77.0] | 25.88 [5.0 to 92.0]

59. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 8
Time Frame: as for outcome 15
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). Subjects in the Full Analysis Set (FAS) with data at this time-point are included. Data collected after receipt of rescue therapy have been set to missing in that study. [Week 8 is the start of Study C87047].
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
mg/L | 23.80 [6.0 to 67.0] | 19.11 [1.0 to 115.0] | 11.61 [5.0 to 67.0]

60. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 12
Time Frame: as for outcome 16
Population: as for outcome 58
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
mg/L | 12.55 [1.0 to 38.0] | 14.91 [1.0 to 100.0] | 11.64 [4.0 to 56.0]

61. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 16
Time Frame: as for outcome 17
Population: as for outcome 58
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
mg/L | 16.12 [1.0 to 58.0] | 16.06 [1.0 to 99.0] | 14.05 [5.0 to 76.0]

62. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 20
Time Frame: as for outcome 18
Population: as for outcome 58
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
mg/L | 17.16 [0.0 to 47.0] | 13.16 [3.0 to 73.0] | 17.44 [4.0 to 63.0]

63. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 24
Time Frame: as for outcome 19
Population: as for outcome 58
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
mg/L | 10.97 [1.0 to 40.0] | 12.44 [1.0 to 77.0] | 16.84 [5.0 to 87.0]

64. Secondary Outcome: C-Reactive Protein (CRP) Level at Week 26
Time Frame: as for outcome 20
Population: as for outcome 58
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
mg/L | 15.94 [0.0 to 48.0] | 9.96 [2.0 to 43.0] | 13.11 [4.0 to 78.0]

65. Secondary Outcome: C-Reactive Protein (CRP) Level at Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals)
Time Frame: as for outcome 21
Population: as for outcome 58
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
mg/L | 19.81 [0.0 to 48.0] | 13.12 [2.0 to 81.0] | 14.04 [4.0 to 78.0]

66. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 8 to Week 0
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
ratio | 1.11 [0.5 to 6.0] | 0.73 [0.1 to 5.6] | 0.45 [0.1 to 1.4]

67. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 12 to Week 0
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 14 | 15
ratio | 0.63 [0.2 to 1.4] | 0.55 [0.1 to 1.7] | 0.45 [0.1 to 1.4]

68. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 16 to Week 0
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 8 | 13 | 14
ratio | 0.81 [0.2 to 1.9] | 0.59 [0.1 to 1.9] | 0.53 [0.3 to 2.4]

69. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 20 to Week 0
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 12 | 14
ratio | 0.65 [0.0 to 1.4] | 0.53 [0.1 to 1.9] | 0.66 [0.1 to 2.0]

70. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 24 to Week 0
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 6 | 11 | 13
ratio | 0.72 [0.2 to 1.8] | 0.5 [0.1 to 1.7] | 0.62 [0.1 to 1.8]

71. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Week 26 to Week 0
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 5 | 11 | 12
ratio | 0.63 [0.0 to 1.2] | 0.4 [0.1 to 1.7] | 0.47 [0.1 to 2.5]

72. Secondary Outcome: Ratio of C-Reactive Protein (CRP) Level at Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) to Week 0
Time Frame: as for outcome 8
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 7 | 13 | 13
ratio | 0.72 [0.0 to 1.2] | 0.48 [0.1 to 1.8] | 0.52 [0.1 to 2.5]

73. Secondary Outcome: Percentage of Subjects at Week 8 Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Responders at Week 6 of double-blind main study, C87037 (NCT00291668) could enter this open-label extension study, C87047 (NCT00329550). All subjects in the Full Analysis Set (FAS) were included in this summary. If a subject withdrew or received rescue therapy, they were counted as a non-responder in that study from that time-point onwards.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 77.8 | 73.3 | 86.7
  Percentage of 70-point non-responders | 22.2 | 26.7 | 13.3

74. Secondary Outcome: Percentage of Subjects at Week 12 Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 73
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 77.8 | 80.0 | 93.3
  Percentage of 70-point non-responders | 22.2 | 20.0 | 6.7

75. Secondary Outcome: Percentage of Subjects at Week 16 Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 73
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 77.8 | 66.7 | 66.7
  Percentage of 70-point non-responders | 22.2 | 33.3 | 33.3

76. Secondary Outcome: Percentage of Subjects at Week 20 Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 5
Population: as for outcome 73
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 66.7 | 60.0 | 73.3
  Percentage of 70-point non-responders | 33.3 | 40.0 | 26.7

77. Secondary Outcome: Percentage of Subjects at Week 24 Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 6
Population: as for outcome 73
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 55.6 | 66.7 | 60.0
  Percentage of 70-point non-responders | 44.4 | 33.3 | 40.0

78. Secondary Outcome: Percentage of Subjects at Week 26 Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 73
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 55.6 | 73.3 | 73.3
  Percentage of 70-point non-responders | 44.4 | 26.7 | 26.7

79. Secondary Outcome: Percentage of Subjects at Last Visit (Week 26 for Completers or the Withdrawal Visit for Premature Withdrawals) Achieving a Reduction in Crohn's Disease Activity Index (CDAI) Score of ≥70 Points From Week 0
Description: as for outcome 2
Time Frame: as for outcome 8
Population: as for outcome 73
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
Percentage of subjects
  Percentage of 70-point responders | 55.6 | 73.3 | 73.3
  Percentage of 70-point non-responders | 44.4 | 26.7 | 26.7

80. Post Hoc Outcome: Number of Subjects With Disease Progression
Description: Disease progression is defined as:
  * an increase from Week 6 of ≥100 points in Crohn's Disease Activity Index (CDAI) score and CDAI >175 points for at least 2 consecutive visits,
  * use of rescue therapy, or,
  * subject withdrawal from the study.
Time Frame: as for outcome 22
Population: Responders at Week 6 of Study C87037 (NCT00291668) could enter this extension study, C87047 (NCT00329550). As it was not possible to calculate the time to disease progression (outcome measure 22) due to the very small number of subjects meeting this definition, the post-hoc outcome of number of subjects with disease progression is presented here.
Measure: Number; unit: subjects
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg
Number analyzed (Participants) | 9 | 15 | 15
subjects | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data summarized in the first four columns were collected from the day after the end of the double-blind main study up to and including 12 weeks following the last dose received in this extension study for each subject (i.e., up to 30 weeks).
Description: For the fifth column, 'Total 2', this presents the data summarized in 'Total 1' PLUS adverse event data from the double-blind main study for subjects who received certolizumab pegol (CZP) in the main study and then entered this extension study (i.e., up to 36 weeks).
Groups:
- Total 1 (This Extension Study Only): This includes all adverse event data collected in this extension study for all 40 subjects who entered this extension study.
- Total 2 (Treatment With CZP in Main Study and Extension Study): This includes all adverse event data from the 6-week double-blind main study (NCT00291668) and this extension study for all 40 subjects who entered this extension study, whilst they were receiving treatment with certolizumab pegol (CZP) in either study. Adverse events recorded in the double-blind main study (NCT00291668) for subjects who received Placebo treatment during that study are not included here.
Arm/Group | CZP 400 mg / Placebo | CZP 400 mg / CZP 200 mg | CZP 400 mg / CZP 400 mg | Total 1 (This Extension Study Only) | Total 2 (Treatment With CZP in Main Study and Extension Study)
Serious Adverse Events (participants affected / at risk) | 2/9 | 5/15 | 5/16 | 12/40 | 13/40
Other Adverse Events (participants affected / at risk) | 8/9 | 12/15 | 15/16 | 35/40 | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 400 mg / Placebo (N=9) | CZP 400 mg / CZP 200 mg (N=15) | CZP 400 mg / CZP 400 mg (N=16) | Total 1 (This Extension Study Only) (N=40) | Total 2 (Treatment With CZP in Main Study and Extension Study) (N=40)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 8 (8) | 8 (8)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP 400 mg / Placebo (N=9) | CZP 400 mg / CZP 200 mg (N=15) | CZP 400 mg / CZP 400 mg (N=16) | Total 1 (This Extension Study Only) (N=40) | Total 2 (Treatment With CZP in Main Study and Extension Study) (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Antinuclear antibody increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Antinuclear antibody positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis pseudomembranous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
DNA antibody positive (Investigations) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 5 (5)
Dental caries (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Laryngopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4) | 3 (4) | 10 (12) | 15 (20) | 18 (27)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 6 (6)
Neurosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharynx discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (4) | 3 (4)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)

LIMITATIONS AND CAVEATS:
Due to the small number of subjects in this study, the percentages of subjects with adverse events may be misleading.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.